CLINICAL TRIAL: NCT04681963
Title: Clinical Characteristics of Hospitalized Adults With Community-acquired- Pneumonia at the Emergency Department: A Cross-sectional Study
Brief Title: Clinical Characteristics of Acutely Hospitalized Adults With Community-acquired- Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-11e-2020
Record Dates: First submitted 2020-11-23; First posted 2020-12-23 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pneumonia
Keywords: risk factors; Community acquired pneumonia
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected pneumonia diagnosis: Acutely admitted patients suspected having pneumonia.
  Interventions: Other: Clinical Assessment within 4 hours of admission

INTERVENTIONS:
Other: Clinical Assessment within 4 hours of admission — Demographics, Symptoms, Severity scores (Triage at admission, confusion, urea, respiration, blood pressure, age (CURB 65) and pneumonia severity score (PSI), clinical parameters, blood testing, chest x-rays, comorbidities, electro-cardiogram

SUMMARY:
There is no gold standard when diagnosing of pneumonia. The variability of clinical signs and symptoms make it difficult to distinguish pneumonia from other causes of respiratory conditions. Well defined characteristics upon arrival to the emergency department will contribute to the better and quicker diagnosis of community-acquired pneumonia.

DETAILED DESCRIPTION:
Currently, pneumonia diagnosis is primarily based on clinical symptoms such as cough, shortness of breath, chest pain, fever and sputum production, combined with X-ray of the lungs, relevant blood tests and microbiological analysis of sputum samples. The X-ray is an imprecise diagnostic tool, and results from sputum assays are first available after 2 days. In the elderly, pneumonia presents with clinically differing signs such as delirium, malnutrition, and there may be an absence of fever, cough and dyspnea. The physical examination is also challenged by a broad variety of atypical symptoms like headache, dry cough and gastrointestinal symptoms in the form of nausea, vomiting or diarrhea. Our hypothesis is that well-defined clinical characteristics upon arrival to the emergency department will contribute to the better and quicker diagnosis of pneumonia.

The aim is to identify the information available upon arrival to the Emergency Department that contributes to diagnosis and prognosis of community-acquired-pneumonia.

The objectives are:

1. Identify the information available upon arrival that correlates to the diagnosis of community-acquired pneumonia
2. Identify the information available upon arrival that correlates to severity of community-acquired pneumonia

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patients suspected with CAP by the attending physician. The physician will base his/her suspicion on e.g. clinical symptoms such as cough, increased sputum production, chest tights, dyspnea and fever>38C, and indication for x-ray.

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients suspected of community-acquired pneumonia at three hospitals in The Region of Southern Denmark (Hospital Sønderjylland, Hospital Lillebaelt and Odense University Hospital).
Sampling Method: Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of community acquired pneumonia | expert assessment within 3 months after patient discharge from the hospital
  The percentage of patients diagnosed with community-acquired pneumonia determined by an expert panel. This outcome measure is a binary variable - verified pneumonia or no pneumonia.
  The expert panel consists of two independent consultants from the emergency department with experience in infection and emergency medicine, who individually will determine whether or not the patient admitted with suspected community-acquired pneumonia had the diagnosis. The diagnosis will be based on all available relevant information from the patient medical record within 48 hours from admission including computed tomography. A standardized template will be used. Disagreement will be discussed until a consensus is reached.

SECONDARY OUTCOMES:
Intensive care unit (ICU) treatment: | within 60 days from admission to the emergency department
  Transfer to the intensive care unit will be recorded during the current hospitalization as a binary variable (transferred/not-transferred)
Length of hospital stay | within 60 days from current admission to the emergency department
  Defined as the time (in days) spent in hospital during the current admission. Measured in days from admission to hospital discharge. Discharge date minus admission date
30-days mortality | 30 days from the admission to the emergency department
  Mortality within 30 days from admission to the Emergency Department
Readmission | within 30 days from the discharge to the hospital
  If a subject is admitted over a 30 day period after the current hospitalization discharge measured as a binary outcome Re-admissions/not re-admissions.
In-hospital mortality | within 60 days from admission to the emergency department
  Patient mortality during the current hospitalization. Binary outcome - Died/ Not died

OTHER OUTCOMES:
90 days mortality | within 90 days from admission to emergency department
  binary
CURB-65 score for predicting mortality in community-acquired-pneumonia | within 4 hours from admission
  CURB-65 score consists of: Confusion of new onset, Blood Urea nitrogen greater than 7 mmol/L (19 mg/dL), respiratory rate of 30 breaths per minute or greater, blood pressure less than 90 mmHg systolic or diastolic blood pressure 60 mmHg or less and age 65 or older. The score stratify patients to groups 1 (mild pneumonia), 2 (moderate pneumonia) and 3-5 (severe pneumonia).
Pneumonia severity index (PSI) | : within 4 hours from admission
  Risk classes to predict the severity of pneumonia. Scores are given based on demographics, comorbidity, clinical measurements and physical Exam Findings (<70 = Risk Class II, 71-90 = Risk Class III, 91-130 = Risk Class IV, >130 = Risk Class V)
Microbial agents | results within 7 days from sputum sample collection
  Microbial agents (bacteria and viruses) identified in standard culture, PCR and multiplex PCR. Sputum samples are collected within 1 hour from patient admission. Descriptive findings in percentage will be registered.
Level of infection markers | results within 4 hour from admission
  Concentration of serum PCT and suPAR are collected in connection to routine blood tests within 1 hour from admission.
Level of markers of lung injury | within 4 hours from admission
  Concentration of serum surfactant protein D, KL-6 and YKL-40
Bacteriuria | within 4 hours from admission
  Binary outcome defined by the microbiologist on urine culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres A, Blasi F, Peetermans WE, Viegi G, Welte T. The aetiology and antibiotic management of community-acquired pneumonia in adults in Europe: a literature review. Eur J Clin Microbiol Infect Dis. 2014 Jul;33(7):1065-79. doi: 10.1007/s10096-014-2067-1. Epub 2014 Feb 15. PMID 24532008
- [Background] Marti C, Garin N, Grosgurin O, Poncet A, Combescure C, Carballo S, Perrier A. Prediction of severe community-acquired pneumonia: a systematic review and meta-analysis. Crit Care. 2012 Jul 27;16(4):R141. doi: 10.1186/cc11447. PMID 22839689
- [Background] Musher DM, Roig IL, Cazares G, Stager CE, Logan N, Safar H. Can an etiologic agent be identified in adults who are hospitalized for community-acquired pneumonia: results of a one-year study. J Infect. 2013 Jul;67(1):11-8. doi: 10.1016/j.jinf.2013.03.003. Epub 2013 Mar 19. PMID 23523447
- [Background] Garau J, Baquero F, Perez-Trallero E, Perez JL, Martin-Sanchez AM, Garcia-Rey C, Martin-Herrero JE, Dal-Re R; NACER Group. Factors impacting on length of stay and mortality of community-acquired pneumonia. Clin Microbiol Infect. 2008 Apr;14(4):322-9. doi: 10.1111/j.1469-0691.2007.01915.x. Epub 2008 Jan 8. PMID 18190569
- [Background] Metlay JP, Kapoor WN, Fine MJ. Does this patient have community-acquired pneumonia? Diagnosing pneumonia by history and physical examination. JAMA. 1997 Nov 5;278(17):1440-5. PMID 9356004
- [Background] McLaughlin JM, Khan FL, Thoburn EA, Isturiz RE, Swerdlow DL. Rates of hospitalization for community-acquired pneumonia among US adults: A systematic review. Vaccine. 2020 Jan 22;38(4):741-751. doi: 10.1016/j.vaccine.2019.10.101. Epub 2019 Dec 13. PMID 31843272
- [Background] Sogaard M, Nielsen RB, Schonheyder HC, Norgaard M, Thomsen RW. Nationwide trends in pneumonia hospitalization rates and mortality, Denmark 1997-2011. Respir Med. 2014 Aug;108(8):1214-22. doi: 10.1016/j.rmed.2014.05.004. Epub 2014 May 20. PMID 24898129
- [Derived] Skjot-Arkil H, Cartuliares MB, Heltborg A, Lorentzen MH, Hertz MA, Kaldan F, Specht JJ, Graumann O, Lindberg MJH, Mikkelsen PA, Nielsen SL, Jensen J, Roge BT, Rosenvinge FS, Mogensen CB. Clinical characteristics and diagnostic accuracy of preliminary diagnoses in adults with infections in Danish emergency departments: a multicentre combined cross-sectional and diagnostic study. BMJ Open. 2024 Dec 5;14(12):e090259. doi: 10.1136/bmjopen-2024-090259. PMID 39638587
- [Derived] Cartuliares MB, Mogensen CB, Rosenvinge FS, Skovsted TA, Lorentzen MH, Heltborg A, Hertz MA, Kaldan F, Specht JJ, Skjot-Arkil H. Community-acquired pneumonia: use of clinical characteristics of acutely admitted patients for the development of a diagnostic model - a cross-sectional multicentre study. BMJ Open. 2024 May 30;14(5):e079123. doi: 10.1136/bmjopen-2023-079123. PMID 38816044
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497